CLINICAL TRIAL: NCT02415374
Title: Bioavailability and Metabolism of Avenanthramide: a Novel Oat Phytochemical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1314
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Bioavailability; Metabolism; Avenanthramides
MeSH Terms: interventions — avenanthramide-2C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-AVA oat flour cookies (Placebo Comparator): Three low-AVA oat flour cookies
  Interventions: Other: Avenanthramides
- High-AVA oat flour cookies (Experimental): Three high-AVA cookies
  Interventions: Other: Avenanthramides

INTERVENTIONS:
Other: Avenanthramides — AVAs are a group of diphenolic acids that are found only in oats (Avena sativa). In this study, each dietary group of subjects will receive three cookies made with oat flour containing high-AVA (H-AVA, 229.56 mg/kg) and low-AVA (L-AVA, 32.69 mg/kg).

SUMMARY:
The purpose of the study is to examine whether orally ingested oat avenanthramides (AVA) in oat flour cookies are bioavailable in humans by measuring plasma and urine concentrations of AVAs and their potential metabolites after ingestion. The blood and urine concentrations will be quantified at several different time points after the oat flour cookies are consumed to characterize the "concentration-time profile".

ELIGIBILITY:
Inclusion Criteria:

* Male and female non-obese subjects (18kg/M2<BMI<28kg/M2)
* Age 20-45 years)
* Sign an informed consent form approved by UMN-IRB
* Willing to avoid oat consumption and rigorous physical activity the day prior to and through test, and consume a low-flavonoid diet for 1 week prior to the study

Exclusion Criteria:

* Presence of GI conditions that interfere with absorption;
* Clinically significant endocrine, cardiovascular, pulmonary, renal, hepatic, pancreatic, biliary or neurologic disorders;
* Major trauma or surgery within 3 months of visit;
* Cancer in the prior 2 years;
* Allergic to oat products;
* Women who are pregnant or lactating;
* Smoking;
* Drinking alcohol >5 drinks/week;
* Using nutraceuticals;
* Blood pressure medication;
* NSAID (>800 mg ibuprofen/week);
* Vitamin supplementation;
* Anticoagulants or hypoglycemic drugs;
* Oat products consumption the day before the test;
* Rigorous physical activity the day before the test;
* Consumption of a high-flavonoid diet in the week prior to the test.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

PRIMARY OUTCOMES:
iAUC for each AVA | 0-10 hours
Cmax for each AVA | 0-10 hours
Tmax for each AVA | 0-10 hours
T1/2 for each AVA | 0-10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Li Li Ji, PhD, Principal Investigator — School of Kinesiology (Cooke Hall), 1906 University Ave. SE, Minneapolis, MN 55455

REFERENCES:
- [Derived] Zhang T, Shao J, Gao Y, Chen C, Yao D, Chu YF, Johnson J, Kang C, Yeo D, Ji LL. Absorption and Elimination of Oat Avenanthramides in Humans after Acute Consumption of Oat Cookies. Oxid Med Cell Longev. 2017;2017:2056705. doi: 10.1155/2017/2056705. Epub 2017 Dec 21. PMID 29430278